CLINICAL TRIAL: NCT04967183
Title: Polyprev Study: Randomized, Multicenter, Controlled Trial Comparing Fecal Immunochemical Test With Endoscopic Surveillance After Advanced Adenoma Resection in Fecal Immunochemical Test Colorectal Cancer Screening Programs.
Brief Title: Polyprev: Study to Compare Fecal Immunochemical Test With Endoscopic Surveillance After Advanced Adenoma Resection in Fecal Immunochemical Test Colorectal Cancer Screening Programs.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacin Biomedica Galicia Sur (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: POLYPREV
Record Dates: First submitted 2021-07-08; First posted 2021-07-19 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Colorectal Cancer
Keywords: Screening program; Endoscopic surveillance; Fecal immunochemical test; Mediterranean diet; Physical activity
MeSH Terms: conditions — Colorectal Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: Patients will be identified in population CRC secreening programs of Galicia, the Basque Country, the Region of Valencia and Murcia. We will considered individuals aged 50 to 65 years with at least one advanced adenoma (tubulovillous or villous histology, high grade dysplasia or ≥ 10mm), and / or at least three non-advanced adenomas detected and resected completely within the population-based CRC screening program.
  Patients will be randomly allocated to perform an annual FIT and colonoscopy if fecal hemoglobin concentration is ≥10µg/g, or to perform endoscopic surveillance. Patients will be also stratified into two groups: ≥5 adenomas or an adenoma ≥20mm and the rest of patients.
  Patients will be followed for a period of 10 years.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental): Annual FIT surveillance
  Interventions: Diagnostic Test: Annual FIT
- Group II (Active Comparator): Endoscopic surveillance
  Interventions: Procedure: Endoscopic surveillance.

INTERVENTIONS:
Diagnostic Test: Annual FIT — Patients will be offered an annual FIT and colonoscopy will be performed if fecal hemoglobin concentration is ≥10µg / g of feces. After performing a colonoscopy the FIT will be sent to the patient:
  * After one year if the unscheduled colonoscopy has been incomplete or a lesion requiring endoscopic surveillance has been completely resected.
  * After five years if the colonoscopy has evaluated the entire mucosa, it is normal or with lesions that do not require endoscopic surveillance (1-2 non-advanced adenomas).
  Arms: Group I
Procedure: Endoscopic surveillance. — First surveillance colonoscopy will be performed in three-year time. If an advanced adenoma or at least three non-advanced adenomas are detected, colonoscopy will be repeated after 3 years. In contrast, if colonoscopy is normal or 1-2 non-advanced adenomas are detected, colonoscopy will be repeated after 5 years.
  Arms: Group II

SUMMARY:
Colorectal cancer (CRC) screening programs have been implemented to reduce the burden of the disease. When an advanced colonic lesions is detected, it is recommended to perform endoscopic surveillance with different intervals between explorations. Although the reduction in CRC incidence, endoscopic surveillance is producing a considerable increase in the number of colonoscopies. However, participation in CRC screening programs based on the fecal immunochemical test (FIT) could be a non inferior alternative to endoscopic surveillance.

Based on this hypothesis, the research group have designed a randomized clinical trial within the population CRC screening programs to compare FIT surveillance to endoscopic surveillance in patients with advanced lesions resected.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is one of the most common malignancies in western countries. CRC screening programs have been implemented in order to reduce the burden of the disease. Screening programs in Spain are based on the biennial detection of fecal hemoglobin with a fecal immunochemical test (FIT) and a diagnostic colonoscopy if positive. The detection of at least one advanced adenoma or serrated lesion defines a high risk situation for metachronous CRC. This group of patients is recommended to perform endoscopic surveillance with different intervals between explorations. Endoscopic surveillance reduces mortality only 1.7% and increases the number of colonoscopies by 62% with an additional cost of € 68,000 for an increase of 0.9 years of life. Moreover, colonoscopy is a procedure associated with potentially serious side effects.

A recently British study shows that with a cut-off of 10 µg/g, FIT has a higher sensitivity and specificity for CRC with a significant cost reduction compared to colonoscopy surveillance. Additionally, most of the population prefers non-invasive faecal tests rather than colonoscopy.

Based on this evidence, the research group have designed a multicenter, randomized clinical trial to compare the 10 year CRC incidence after resection of advanced colonic lesions detected within CRC screening programs between endoscopic surveillance and participation in CRC screening programs based on FIT.

Apart from this purpose, the investigators will also assess the values and preferences regarding surveillance and risk of CRC. Further, the research group will evaluate the relationship between Mediterranean diet and physical activity with the detection of advanced adenomas and CRC.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged 50 to 65 years.
2. Individuals with at least one advanced adenoma (tubulovillous or villous histology, high grade dysplasia or ≥ 10mm), and / or at least three non-advanced adenomas detected and resected completely within the population-based CRC screening program.

Exclusion Criteria:

1. Personal history of CRC.
2. Colonic lesion ≥10mm resected without histological diagnosis.
3. More than 10 adenomas in baseline colonoscopy.
4. Serrated polyposis syndrome.
5. Two or more first-degree relatives with CRC.
6. Hereditary predisposition to CRC.
7. Relevant comorbidity with life expectancy inferior to 5 years.
8. Colonoscopy with incomplete mucosal examination.
9. Incomplete resection of baseline lesions.
10. Non-acceptance after reading the informed consent.

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3788 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2035-06 (Estimated)

PRIMARY OUTCOMES:
Rate of invasive CRC | 10 years
  It is the main outcome of the study. Invasive CRC is defined as colonic adenocarcinoma that invades the submucosa. Adenocarcinomas in situ and intramucosal carcinomas will not be considered as invasive CRC.
Rate of interval CRC | 10 years
  Interval CRC is defined as the CRC detected between two organized surveillance (FIT or colonoscopy).
Mortality | 10 years
  The deaths and their cause will be collected: associated with CRC, associated with adverse effects of screening or unrelated.
Rate of advanced colonic lesions | 10 years
  Advanced colonic lesions will be defined as advanced adenomas (at least 10mm, hairy histology or high grade dysplasia) or advanced serrated lesions (at least 10mm or with dysplasia).
Frequency of participation in the surveillance strategy | 10 years
  According to the methodology of the information systems of the screening programs, three categories will be defined: non-participation, irregular participation, regular participation.
Adverse effects | 10 years
  Adverse effects associated with surveillance are defined as complications that require hospitalization. Those related to the surgical treatment of benign colonic lesions will be included as adverse effects.

SECONDARY OUTCOMES:
CRC, adenoma and advanced serrated lesions at three years | 3 years
  Detection of CRC, adenoma and advanced serrated lesion will be collected at 3 years of follow-up.
Physical activity | 3 years
  We will use the International Physical Activity. Questionnaire (IPAQ) to mesure physical activity.
Mediterranean lifestyle | 3 years
  We will use the Mediterranean Lifestyle index (MEDLIFE) to measure overall adherence to the Mediterranean lifestyle.
Preferences of the subjects | 2 years
  We will use a survey with vignette questions to evaluate the values and preferences of the subjects regarding surveillance.

CONTACTS AND LOCATIONS:
Locations (1):
- Complexo Hospitalario Universitario de Ourense, Ourense, Spain

REFERENCES:
- [Background] Holleczek B, Rossi S, Domenic A, Innos K, Minicozzi P, Francisci S, Hackl M, Eisemann N, Brenner H; EUROCARE-5 Working Group:. On-going improvement and persistent differences in the survival for patients with colon and rectum cancer across Europe 1999-2007 - Results from the EUROCARE-5 study. Eur J Cancer. 2015 Oct;51(15):2158-2168. doi: 10.1016/j.ejca.2015.07.024. Epub 2015 Sep 26. PMID 26421819
- [Background] Atkin WS, Valori R, Kuipers EJ, Hoff G, Senore C, Segnan N, Jover R, Schmiegel W, Lambert R, Pox C; International Agency for Research on Cancer. European guidelines for quality assurance in colorectal cancer screening and diagnosis. First Edition--Colonoscopic surveillance following adenoma removal. Endoscopy. 2012 Sep;44 Suppl 3:SE151-63. doi: 10.1055/s-0032-1309821. Epub 2012 Sep 25. PMID 23012119
- [Background] Bretthauer M, Loberg M, Kalager M. Long-term colorectal-cancer mortality after adenoma removal. N Engl J Med. 2014 Nov 20;371(21):2036-7. doi: 10.1056/NEJMc1411954. No abstract available. PMID 25409378
- [Background] Zauber AG, Winawer SJ, O'Brien MJ, Lansdorp-Vogelaar I, van Ballegooijen M, Hankey BF, Shi W, Bond JH, Schapiro M, Panish JF, Stewart ET, Waye JD. Colonoscopic polypectomy and long-term prevention of colorectal-cancer deaths. N Engl J Med. 2012 Feb 23;366(8):687-96. doi: 10.1056/NEJMoa1100370. PMID 22356322
- [Background] Martinez ME, Baron JA, Lieberman DA, Schatzkin A, Lanza E, Winawer SJ, Zauber AG, Jiang R, Ahnen DJ, Bond JH, Church TR, Robertson DJ, Smith-Warner SA, Jacobs ET, Alberts DS, Greenberg ER. A pooled analysis of advanced colorectal neoplasia diagnoses after colonoscopic polypectomy. Gastroenterology. 2009 Mar;136(3):832-41. doi: 10.1053/j.gastro.2008.12.007. Epub 2008 Dec 9. PMID 19171141
- [Background] Hassan C, Quintero E, Dumonceau JM, Regula J, Brandao C, Chaussade S, Dekker E, Dinis-Ribeiro M, Ferlitsch M, Gimeno-Garcia A, Hazewinkel Y, Jover R, Kalager M, Loberg M, Pox C, Rembacken B, Lieberman D; European Society of Gastrointestinal Endoscopy. Post-polypectomy colonoscopy surveillance: European Society of Gastrointestinal Endoscopy (ESGE) Guideline. Endoscopy. 2013 Oct;45(10):842-51. doi: 10.1055/s-0033-1344548. Epub 2013 Sep 12. PMID 24030244
- [Background] Cubiella J, Carballo F, Portillo I, Cruzado Quevedo J, Salas D, Binefa G, Mila N, Hernandez C, Andreu M, Teran A, Arana-Arri E, Ono A, Valverde MJ, Bujanda L, Hernandez V, Morillas JD, Jover R, Castells A. Incidence of advanced neoplasia during surveillance in high- and intermediate-risk groups of the European colorectal cancer screening guidelines. Endoscopy. 2016 Nov;48(11):995-1002. doi: 10.1055/s-0042-112571. Epub 2016 Aug 2. PMID 27485482
- [Background] Mangas-Sanjuan C, Jover R, Cubiella J, Marzo-Castillejo M, Balaguer F, Bessa X, Bujanda L, Bustamante M, Castells A, Diaz-Tasende J, Diez-Redondo P, Herraiz M, Mascort-Roca JJ, Pellise M, Quintero E; Grupo de Cribado del Cancer Colorrectal de la Sociedad Espanola de Epidemiologia. Endoscopic surveillance after colonic polyps and colorrectal cancer resection. 2018 update. Gastroenterol Hepatol. 2019 Mar;42(3):188-201. doi: 10.1016/j.gastrohep.2018.11.001. Epub 2019 Jan 6. English, Spanish. PMID 30621911
- [Background] Zorzi M, Senore C, Turrin A, Mantellini P, Visioli CB, Naldoni C, Sassoli De' Bianchi P, Fedato C, Anghinoni E, Zappa M, Hassan C; Italian colorectal cancer screening survey group. Appropriateness of endoscopic surveillance recommendations in organised colorectal cancer screening programmes based on the faecal immunochemical test. Gut. 2016 Nov;65(11):1822-1828. doi: 10.1136/gutjnl-2015-310139. Epub 2015 Aug 21. PMID 26297727
- [Background] Lieberman DA, Holub J, Eisen G, Kraemer D, Morris CD. Utilization of colonoscopy in the United States: results from a national consortium. Gastrointest Endosc. 2005 Dec;62(6):875-83. doi: 10.1016/j.gie.2005.06.037. PMID 16301030
- [Background] Marzo-Castillejo M, Almeda J, Mascort JJ, Cunillera O, Saladich R, Nieto R, Pineiro P, Llagostera M, Cantero F, Segarra M, Puente D. Appropriateness of colonoscopy requests according to EPAGE-II in the Spanish region of Catalonia. BMC Fam Pract. 2015 Oct 26;16:154. doi: 10.1186/s12875-015-0369-8. PMID 26498043
- [Background] Greuter MJE, de Klerk CM, Meijer GA, Dekker E, Coupe VMH. Screening for Colorectal Cancer With Fecal Immunochemical Testing With and Without Postpolypectomy Surveillance Colonoscopy: A Cost-Effectiveness Analysis. Ann Intern Med. 2017 Oct 17;167(8):544-554. doi: 10.7326/M16-2891. Epub 2017 Oct 3. PMID 28973514
- [Background] Atkin W, Cross AJ, Kralj-Hans I, MacRae E, Piggott C, Pearson S, Wooldrage K, Brown J, Lucas F, Prendergast A, Marchevsky N, Patel B, Pack K, Howe R, Skrobanski H, Kerrison R, Swart N, Snowball J, Duffy SW, Morris S, von Wagner C, Halloran S. Faecal immunochemical tests versus colonoscopy for post-polypectomy surveillance: an accuracy, acceptability and economic study. Health Technol Assess. 2019 Jan;23(1):1-84. doi: 10.3310/hta23010. PMID 30618357
- [Background] Bonello B, Ghanouni A, Bowyer HL, MacRae E, Atkin W, Halloran SP, Wardle J, von Wagner C. Using a hypothetical scenario to assess public preferences for colorectal surveillance following screening-detected, intermediate-risk adenomas: annual home-based stool test vs. triennial colonoscopy. BMC Gastroenterol. 2016 Sep 13;16(1):113. doi: 10.1186/s12876-016-0517-1. PMID 27618798
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Sotos-Prieto M, Moreno-Franco B, Ordovas JM, Leon M, Casasnovas JA, Penalvo JL. Design and development of an instrument to measure overall lifestyle habits for epidemiological research: the Mediterranean Lifestyle (MEDLIFE) index. Public Health Nutr. 2015 Apr;18(6):959-67. doi: 10.1017/S1368980014001360. Epub 2014 Jul 15. PMID 25025396
- See also: Related Info — https://redecan.org/redecan.org/es/444_Estimaciones_Incidencia_y_Supervi_Cancer_en_Espa_na_2014_DEF_DEF3a26.pdf?file=257&area=196